CLINICAL TRIAL: NCT03198767
Title: A Randomized, Open Label, Two-part, Three-period, Cross Over Study to Investigate the Effects of Carbohydrate in Diet and to Evaluate Supplements on the Gastrointestinal Tolerability of LIK066 in Overweight or Obese Subjects
Brief Title: Effects of Carbohydrate in Diet and Supplements on the Gastrointestinal Tolerability of LIK066
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CLIK066B2203
Record Dates: First submitted 2017-06-16; First posted 2017-06-26 (Actual); Results first posted 2018-09-25 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-05

CONDITIONS: Obesity
Keywords: obesity; overweight; body mass index; BMI; diarrhea
MeSH Terms: conditions — Obesity; Overweight; Diarrhea | interventions — licogliflozin; Psyllium; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A: LIK066 + P1: 50% CHO / P2: 25% CHO / P3: 0% CHO (Experimental): Period 1 (Day 1-3): Daily dose of 50 mg LIK066 + 50% carbohydrate (CHO) Period 2 (Day 9-11): Daily dose of 50 mg LIK066 + 25% carbohydrate Period 3 (Day 17-19): Daily dose of 50 mg LIK066 + 0% carbohydrate
  Interventions: Drug: LIK066; Dietary Supplement: Carbohydrate 50%; Dietary Supplement: Carbohydrate 25%; Dietary Supplement: Carbohydrate 0%
- Part A: LIK066 + P1: 25% CHO / P2: 0% CHO / P3: 50% CHO (Experimental): Period 1 (Day 1-3): Daily dose of 50 mg LIK066 + 25% carbohydrate (CHO) Period 2 (Day 9-11): Daily dose of 50 mg LIK066 + 0% carbohydrate Period 3 (Day 17-19): Daily dose of 50 mg LIK066 + 50% carbohydrate
  Interventions: Drug: LIK066; Dietary Supplement: Carbohydrate 50%; Dietary Supplement: Carbohydrate 25%; Dietary Supplement: Carbohydrate 0%
- Part A: LIK066 + P1: 0% CHO / P2: 50% CHO / P3: 25% CHO (Experimental): Period 1 (Day 1-3): Daily dose of 50 mg LIK066 + 0% carbohydrate (CHO) Period 2 (Day 9-11): Daily dose of 50 mg LIK066 + 50% carbohydrate Period 3 (Day 17-19): Daily dose of 50 mg LIK066 + 25% carbohydrate
  Interventions: Drug: LIK066; Dietary Supplement: Carbohydrate 50%; Dietary Supplement: Carbohydrate 25%; Dietary Supplement: Carbohydrate 0%
- Part A: LIK066 + P1: 8% CHO (Experimental): Period 1 (Day 1-3): Daily dose of 50 mg LIK066 + 8% carbohydrate (CHO) PROTOCOL DEVIATION: subjects received 8% CHO in error and were discontinued after Period 1.
  Interventions: Drug: LIK066; Dietary Supplement: Carbohydrate 8%
- Part B: LIK066 + 50% CHO + P1: NS / P2: PS / P3: CC (Experimental): Period 1 (Day 1-3): Daily dose of 50 mg LIK066+50% carbohydrate + no supplement (NS) Period 2 (Day 9-11): Daily dose of 50 mg LIK066+50% carbohydrate + 6 g psyllium (PS) Period 3 (Day 17-19): Daily dose of 50 mg LIK066+50% carbohydrate +1g calcium carbonate (CC)
  Interventions: Drug: LIK066; Dietary Supplement: Carbohydrate 50%; Dietary Supplement: Psyllium; Dietary Supplement: Calcium carbonate
- Part B: LIK066 + 50% CHO + P1: PS / P2: CC / P3: NS (Experimental): Period 1 (Day 1-3): Daily dose of 50 mg LIK066+50% carbohydrate + 6 g psyllium (PS) Period 2 (Day 9-11): Daily dose of 50 mg LIK066+50% carbohydrate +1g calcium carbonate (CC) Period 3 (Day 17-19): Daily dose of 50 mg LIK066+50% carbohydrate + no supplement (NS)
  Interventions: Drug: LIK066; Dietary Supplement: Carbohydrate 50%; Dietary Supplement: Psyllium; Dietary Supplement: Calcium carbonate
- Part B: LIK066 + 50% CHO + P1: CC / P2: NS / P3: PS (Experimental): Period 1 (Day 1-3): Daily dose of 50 mg LIK066+50% carbohydrate +1g calcium carbonate (CC) Period 2 (Day 9-11): Daily dose of 50 mg LIK066+50% carbohydrate + no supplement (NS) Period 3 (Day 17-19): Daily dose of 50 mg LIK066+50% carbohydrate + 6 g psyllium (PS)
  Interventions: Drug: LIK066; Dietary Supplement: Carbohydrate 50%; Dietary Supplement: Psyllium; Dietary Supplement: Calcium carbonate

INTERVENTIONS:
Drug: LIK066 — LIK066 50 mg tablets. Open-label, bulk, blister-pack.
Dietary Supplement: Carbohydrate 50% — 50% carbohydrate in breakfast meal
  Arms: Part A: LIK066 + P1: 0% CHO / P2: 50% CHO / P3: 25% CHO; Part A: LIK066 + P1: 25% CHO / P2: 0% CHO / P3: 50% CHO; Part A: LIK066 + P1: 50% CHO / P2: 25% CHO / P3: 0% CHO; Part B: LIK066 + 50% CHO + P1: CC / P2: NS / P3: PS; Part B: LIK066 + 50% CHO + P1: NS / P2: PS / P3: CC; Part B: LIK066 + 50% CHO + P1: PS / P2: CC / P3: NS
Dietary Supplement: Carbohydrate 25% — 25% carbohydrate in breakfast meal
  Arms: Part A: LIK066 + P1: 0% CHO / P2: 50% CHO / P3: 25% CHO; Part A: LIK066 + P1: 25% CHO / P2: 0% CHO / P3: 50% CHO; Part A: LIK066 + P1: 50% CHO / P2: 25% CHO / P3: 0% CHO
Dietary Supplement: Carbohydrate 8% — 8% carbohydrate in breakfast meal
  Arms: Part A: LIK066 + P1: 8% CHO
Dietary Supplement: Carbohydrate 0% — 0% carbohydrate in breakfast meal
  Arms: Part A: LIK066 + P1: 0% CHO / P2: 50% CHO / P3: 25% CHO; Part A: LIK066 + P1: 25% CHO / P2: 0% CHO / P3: 50% CHO; Part A: LIK066 + P1: 50% CHO / P2: 25% CHO / P3: 0% CHO
Dietary Supplement: Psyllium — Powder 6 grams
  Other Names: MetaMucil®
  Arms: Part B: LIK066 + 50% CHO + P1: CC / P2: NS / P3: PS; Part B: LIK066 + 50% CHO + P1: NS / P2: PS / P3: CC; Part B: LIK066 + 50% CHO + P1: PS / P2: CC / P3: NS
Dietary Supplement: Calcium carbonate — Liquid 1 gram (4 mL equivalent sugar free)
  Other Names: Quality Value®
  Arms: Part B: LIK066 + 50% CHO + P1: CC / P2: NS / P3: PS; Part B: LIK066 + 50% CHO + P1: NS / P2: PS / P3: CC; Part B: LIK066 + 50% CHO + P1: PS / P2: CC / P3: NS

SUMMARY:
The purpose of this study was to determine if LIK066 taken with a meal containing low carbohydrate is associated with less diarrhea compared to a high carbohydrate meal and to assess the potential effects of supplements such as psyllium or calcium carbonate on alleviating diarrhea associated with LIK066.

ELIGIBILITY:
Inclusion Criteria:

* obese and overweight, BMI 25-50, HbA1C <10%

Exclusion Criteria:

* Preexisting, clinically significant cardiovascular, liver, renal, or GI disease that is considered unstable; pregnancy, Type 1 diabetes; Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2017-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=453

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 116 subjects were screened and 54 subjects were enrolled and randomized, with 48 completing the study. 6 subjects in Part A were discontinued due to a protocol deviation after day 3 dosing (the protein drink provided to subjects was incorrect and included 8% carbohydrate).
Period: Overall Study
Arm/Group | Part A: LIK066 + P1: 50% CHO / P2: 25% CHO / P3: 0% CHO | Part A: LIK066 + P1: 25% CHO / P2: 0% CHO / P3: 50% CHO | Part A: LIK066 + P1: 0% CHO / P2: 50% CHO / P3: 25% CHO | Part A: LIK066 + P1: 8% CHO | Part B: LIK066 + 50% CHO + P1: NS / P2: PS / P3: CC | Part B: LIK066 + 50% CHO + P1: PS / P2: CC / P3: NS | Part B: LIK066 + 50% CHO + P1: CC / P2: NS / P3: PS
Started | 8 | 8 | 8 | 6 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 0 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 6 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 6 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set. All subjects that received any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: LIK066 + P1: 50% CHO / P2: 25% CHO / P3: 0% CHO | Part A: LIK066 + P1: 25% CHO / P2: 0% CHO / P3: 50% CHO | Part A: LIK066 + P1: 0% CHO / P2: 50% CHO / P3: 25% CHO | Part A: LIK066 + P1: 8% CHO | Part B: LIK066 + 50% CHO + P1: NS / P2: PS / P3: CC | Part B: LIK066 + 50% CHO + P1: PS / P2: CC / P3: NS | Part B: LIK066 + 50% CHO + P1: CC / P2: NS / P3: PS | Total
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 8 | 8 | 8 | 54
Age, Continuous [Mean (Full Range); unit: Years] — Population: Safety Analysis Set
  Years | 32.1 [21 to 46] | 45.5 [27 to 61] | 43.9 [26 to 63] | 53.3 [51 to 57] | 43.8 [27 to 56] | 50.1 [36 to 62] | 43.3 [29 to 58] | 44.3 [21 to 63]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Safety Analysis Set
  Participants
    Female | 5 | 2 | 2 | 1 | 0 | 3 | 4 | 17
    Male | 3 | 6 | 6 | 5 | 8 | 5 | 4 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Safety Analysis Set
  Participants
    Hispanic or Latino | 3 | 1 | 1 | 0 | 2 | 1 | 0 | 8
    Not Hispanic or Latino | 5 | 7 | 7 | 6 | 6 | 7 | 8 | 46
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Episodes of Diarrhea (Part A and Part B)
Description: Episodes of diarrhea is defined as the total number of stools with a Bristol Stool Chart (BSC) Score of 6 or 7 on day 3 of each treatment period. BSC is frequently used as a measure of consistency, and a score of 6 or 7 (pourable or watery stool) is considered abnormal.
Time Frame: 24 hours on Day 3 of each treatment period
Population: PD Analysis Set. All subjects with any available pharmacodynamic (PD) data and no major protocol deviations with impact on PD data.
Measure: Mean (Standard Deviation); unit: Number of stools
Groups:
- Part A: LIK066 + 50% CHO: Part A: LIK066 + 50% carbohydrate CHO
- Part A: LIK066 + 25% CHO: Part A: LIK066 + 25% carbohydrate CHO
- Part A: LIK066 + 0% CHO: Part A: LIK066 + 0% carbohydrate CHO
- Part B: LIK066 + 50% CHO + NS: Daily dose of 50 mg LIK066+50% carbohydrate + no supplement (NS)
- Part B: LIK066 + 50% CHO + PS: Daily dose of 50 mg LIK066+50% carbohydrate + 6 g psyllium (PS)
- Part B: LIK066 + 50% CHO CC: Daily dose of 50 mg LIK066+50% carbohydrate +1g calcium carbonate (CC)
Arm/Group | Part A: LIK066 + 50% CHO | Part A: LIK066 + 25% CHO | Part A: LIK066 + 0% CHO | Part B: LIK066 + 50% CHO + NS | Part B: LIK066 + 50% CHO + PS | Part B: LIK066 + 50% CHO CC
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
Number of stools | 1.67 (1.74) | 1.25 (1.42) | 0.38 (0.71) | 1.88 (1.51) | 1.46 (1.41) | 1.46 (1.67)
Statistical Analysis 1: Comparison: Part A: LIK066 + 50% CHO vs Part A: LIK066 + 25% CHO; Day 3; Test type: Superiority; p = 0.202, Mixed Models Analysis; Ratio of number of events = 0.71, 80% CI 2-sided [0.50 to 1.00]
Statistical Analysis 2: Comparison: Part A: LIK066 + 50% CHO vs Part A: LIK066 + 0% CHO; Day 3; Test type: Superiority; p < 0.001, Mixed Models Analysis; Ratio of number of events = 0.21, 80% CI 2-sided [0.14 to 0.32]
Statistical Analysis 3: Comparison: Part A: LIK066 + 25% CHO vs Part A: LIK066 + 0% CHO; Day 3; Test type: Superiority; p < 0.001, Mixed Models Analysis; Ratio of number of events = 0.30, 80% CI 2-sided [0.19 to 0.46]
Statistical Analysis 4: Comparison: Part B: LIK066 + 50% CHO + NS vs Part B: LIK066 + 50% CHO + PS; Day 3; Test type: Superiority; p = 0.275, Mixed Models Analysis; Ratio of number of events = 0.79, 80% CI 2-sided [0.60 to 1.04]
Statistical Analysis 5: Comparison: Part B: LIK066 + 50% CHO + NS vs Part B: LIK066 + 50% CHO CC; Day 3; Test type: Superiority; p = 0.234, Mixed Models Analysis; Ratio of number of events = 0.78, 80% CI 2-sided [0.59 to 1.02]
Statistical Analysis 6: Comparison: Part B: LIK066 + 50% CHO + PS vs Part B: LIK066 + 50% CHO CC; Day 3; Test type: Superiority; p = 0.921, Mixed Models Analysis; Ratio of number of events = 0.98, 80% CI 2-sided [0.73 to 1.30]

2. Secondary Outcome: Three-day Total Number of Episodes of Diarrhea (Part A and Part B)
Description: Episodes of diarrhea is defined as the total number of stools with a Bristol Stool Chart (BSC) Score of 6 or 7 on days 1 to 3 of each treatment period. BSC is frequently used as a measure of consistency, and a score of 6 or 7 (pourable or watery stool) is considered abnormal.
Time Frame: Day 1 to 3 of each treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of stools
Arm/Group | Part A: LIK066 + 50% CHO | Part A: LIK066 + 25% CHO | Part A: LIK066 + 0% CHO | Part B: LIK066 + 50% CHO + NS | Part B: LIK066 + 50% CHO + PS | Part B: LIK066 + 50% CHO CC
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
Number of stools | 3.96 (3.01) | 2.83 (2.97) | 1.50 (2.02) | 4.42 (3.41) | 3.46 (3.24) | 4.00 (3.11)
Statistical Analysis 1: Comparison: Part A: LIK066 + 50% CHO vs Part A: LIK066 + 25% CHO; Test type: Superiority; p = 0.040, Mixed Models Analysis; Ratio of number of events = 0.68, 80% CI 2-sided [0.54 to 0.86]
Statistical Analysis 2: Comparison: Part A: LIK066 + 50% CHO vs Part A: LIK066 + 0% CHO; Test type: Superiority; p < 0.001, Mixed Models Analysis; Ratio of number of events = 0.37, 80% CI 2-sided [0.28 to 0.49]
Statistical Analysis 3: Comparison: Part A: LIK066 + 25% CHO vs Part A: LIK066 + 0% CHO; Test type: Superiority; p = 0.008, Mixed Models Analysis; Ratio of number of events = 0.54, 80% CI 2-sided [0.41 to 0.72]
Statistical Analysis 4: Comparison: Part B: LIK066 + 50% CHO + NS vs Part B: LIK066 + 50% CHO + PS; Test type: Superiority; p = 0.141, Mixed Models Analysis; Ratio of number of events = 0.79, 80% CI 2-sided [0.65 to 0.97]
Statistical Analysis 5: Comparison: Part B: LIK066 + 50% CHO + NS vs Part B: LIK066 + 50% CHO CC; Test type: Superiority; p = 0.510, Mixed Models Analysis; Ratio of number of events = 0.90, 80% CI 2-sided [0.74 to 1.10]
Statistical Analysis 6: Comparison: Part B: LIK066 + 50% CHO + PS vs Part B: LIK066 + 50% CHO CC; Test type: Superiority; p = 0.401, Mixed Models Analysis; Ratio of number of events = 1.14, 80% CI 2-sided [0.93 to 1.41]

3. Secondary Outcome: Average Consistency With Bristol Stool Chart (Part A and Part B)
Description: BSC is frequently used as a measure of consistency, ranging from score 1 (hard lumps) to 7 (watery stool).
Time Frame: 24 hours on Day 3 of each treatment period
Population: PD Analysis Set.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Part A: LIK066 + 50% CHO | Part A: LIK066 + 25% CHO | Part A: LIK066 + 0% CHO | Part B: LIK066 + 50% CHO + NS | Part B: LIK066 + 50% CHO + PS | Part B: LIK066 + 50% CHO CC
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
score | 5.45 (1.24) | 5.42 (1.42) | 4.71 (1.45) | 5.81 (1.07) | 5.52 (0.99) | 5.62 (1.02)
Statistical Analysis 1: Comparison: Part A: LIK066 + 50% CHO vs Part A: LIK066 + 25% CHO; Test type: Superiority; p = 0.426, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 80% CI 2-sided [-0.56 to 0.13]
Statistical Analysis 2: Comparison: Part A: LIK066 + 50% CHO vs Part A: LIK066 + 0% CHO; Test type: Superiority; p = 0.001, Mixed Models Analysis; Median Difference (Final Values) = -1.06, 80% CI 2-sided [-1.46 to -0.67]
Statistical Analysis 3: Comparison: Part A: LIK066 + 25% CHO vs Part A: LIK066 + 0% CHO; Test type: Superiority; p = 0.009, Mixed Models Analysis; Mean Difference (Final Values) = -0.85, 80% CI 2-sided [-1.25 to -0.45]
Statistical Analysis 4: Comparison: Part B: LIK066 + 50% CHO + NS vs Part B: LIK066 + 50% CHO + PS; Test type: Superiority; p = 0.135, Mixed Models Analysis; Mean Difference (Final Values) = -0.37, 80% CI 2-sided [-0.68 to -0.05]
Statistical Analysis 5: Comparison: Part B: LIK066 + 50% CHO + NS vs Part B: LIK066 + 50% CHO CC; Test type: Superiority; p = 0.436, Mixed Models Analysis; Median Difference (Final Values) = -0.19, 80% CI 2-sided [-0.50 to 0.12]
Statistical Analysis 6: Comparison: Part B: LIK066 + 50% CHO + PS vs Part B: LIK066 + 50% CHO CC; Test type: Superiority; p = 0.452, Mixed Models Analysis; Median Difference (Final Values) = 0.18, 80% CI 2-sided [-0.13 to 0.49]

4. Secondary Outcome: Average Stool pH (Part A and Part B)
Description: Average PH of Stool at day 3
Time Frame: 24 hours on Day 3 of each treatment period
Population: PD Analysis Set
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part A: LIK066 + 50% CHO | Part A: LIK066 + 25% CHO | Part A: LIK066 + 0% CHO | Part B: LIK066 + 50% CHO + NS | Part B: LIK066 + 50% CHO + PS | Part B: LIK066 + 50% CHO CC
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
pH | 6.35 (0.44) | 6.50 (0.59) | 6.29 (0.23) | 6.52 (0.59) | 6.79 (0.67) | 6.66 (0.50)

5. Secondary Outcome: Average Stool Weight (Part A and Part B)
Description: 24 hour average stool weight on day 3
Time Frame: 24 hours on Day 3 of each treatment period
Population: PD Analysis Set
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Part A: LIK066 + 50% CHO | Part A: LIK066 + 25% CHO | Part A: LIK066 + 0% CHO | Part B: LIK066 + 50% CHO + NS | Part B: LIK066 + 50% CHO + PS | Part B: LIK066 + 50% CHO CC
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
gram | 136.5 (88.99) | 154.5 (87.11) | 116.7 (65.57) | 145.5 (75.21) | 177.1 (138.1) | 164.3 (108.5)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately22 days.
Groups:
- Part A: LIK066 + 8% CHO: Part A: LIK066 + 8% carbohydrate CHO
Arm/Group | Part A: LIK066 + 50% CHO | Part A: LIK066 + 25% CHO | Part A: LIK066 + 0% CHO | Part A: LIK066 + 8% CHO | Part B: LIK066 + 50% CHO + NS | Part B: LIK066 + 50% CHO + PS | Part B: LIK066 + 50% CHO CC
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/6 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/6 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 21/24 | 19/24 | 19/24 | 5/6 | 21/24 | 19/24 | 22/24
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: LIK066 + 50% CHO (N=24) | Part A: LIK066 + 25% CHO (N=24) | Part A: LIK066 + 0% CHO (N=24) | Part A: LIK066 + 8% CHO (N=6) | Part B: LIK066 + 50% CHO + NS (N=24) | Part B: LIK066 + 50% CHO + PS (N=24) | Part B: LIK066 + 50% CHO CC (N=24)
Diarrhea (Gastrointestinal disorders) | 20 | 17 | 14 | 3 | 20 | 17 | 22
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 3 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2 | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 6 | 1 | 5 | 1 | 0 | 2 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 2 | 2 | 4
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 3
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT03198767/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT03198767/SAP_001.pdf